CLINICAL TRIAL: NCT05729802
Title: The Holographic Standardized Patient: Using Mixed Reality to Reduce Barriers to Crisis
Brief Title: The Holographic Standardized Patient
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3777
Record Dates: First submitted 2023-01-06; First posted 2023-02-15 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Medical Emergencies; Educational Problems; Simulation of Physical Illness
Keywords: Mixed Reality; Augmented Reality; Medical Simulation; Hololens

STUDY DESIGN:
Intervention Model Description: It is a two stage study that will: 1) iteratively develop and usability test the HoloSIM software with acute care medicine specialties at Sunnybrook, and 2) determine if the HoloSIM platform is non-inferior to the current teaching and assessment standard of high-fidelity mannequin-based crisis simulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: HoloSIM (intervention) (Experimental): Training by Mixed Reality Simulation
  Interventions: Device: HoloSIM Software via Hololens 2
- Group B: Mannequin (control) (Active Comparator): Training by Mannequin Based Simulation
  Interventions: Other: Training by Mannequin Based Simulation

INTERVENTIONS:
Device: HoloSIM Software via Hololens 2 — Participants will train via a mixed reality simulated crisis scenario using the HoloSIM software on the Microsoft Hololens 2
  Arms: Group A: HoloSIM (intervention)
Other: Training by Mannequin Based Simulation — Participants will train a via traditional mannequin based medical crisis scenario
  Arms: Group B: Mannequin (control)

SUMMARY:
The current pandemic has revealed in-person simulation training and evaluation is vulnerable to disruption, and alternatives are needed which allow remote evaluation. The recently developed Microsoft Hololens headset device allows interactable holograms to be inserted into a user's workspace (mixed reality) - permitting the augmentation of existing clinical and training spaces with holographic (i.e. virtual) patients via the prototype HoloSIM software. This study is the first known research initiative aiming to demonstrate the feasibility and effectiveness of mixed reality for acute medicine training and assessment at a distance.

Space, time, personnel, pandemic, and cost constraints limit opportunities for high-fidelity simulation exercises for post-graduate trainees at Sunnybrook. By developing and demonstrating the effectiveness of this new training modality, increased simulation exercises will lead to a higher quality education experience, better functioning teams, and better patient outcomes.

DETAILED DESCRIPTION:
The study is the first known research initiative aiming to demonstrate that a mixed reality simulation training and assessment modality can be implemented in different clinical contexts and can improve decision making skills and management in a complex crisis scenario.

The investigators hypothesize that a mixed reality simulation training solution is usable, feasible, and can improve decision making skills and management.

It is a two stage study: 1) iteratively develop and usability test the HoloSIM software with acute care medicine specialties at Sunnybrook, and 2) determine if the HoloSIM platform is non-inferior to the current teaching and assessment standard of high-fidelity mannequin-based crisis simulation.

The understanding is that this will be a first-of-its-kind study that will generate an accessible, easy to administer tool to educate residents and fellows. The presented HoloSIM software will allow teams to practice and assess their responses to a variety of scenarios in clinical environments such as the trauma bay and ICU. This has the potential to improve team function and enhance quality of care across the healthcare system.

Healthcare facilities without expensive simulation centres are unable to participate in high-fidelity medical simulation. Inequities in access to high quality training and professional development have been repeatedly cited as a barrier to retention of rural health care providers. The SHSC simulation centre will adapt this approach and offer training at a distance and medical crisis coaching to rural health care providers utilizing the this mentioned platform. Lastly, all simulation resources developed during the project will be made freely available via the project website. Other institutions internationally may use them to improve their team performance, patient safety, and postgraduate education programs.

ELIGIBILITY:
Inclusion Criteria:

* Resident or fellow level volunteers from acute care postgraduate training programs (Internal Medicine, Emergency Medicine, Anesthesiology, Critical Care Medicine at Sunnybrook Health Sciences Centre

Exclusion Criteria:

* Unwilling to enter the study
* Previous experience with simulator based teaching on anaphylaxis

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Anaphylaxis Checklist of Core Decision Making Steps | 30 days post exposure
  Expert consensus based checklists of critical scenario actions on a mannequin based crisis scenario. Student scenario performance graded from 0 to 45, with higher scores representing a better performance.

SECONDARY OUTCOMES:
System Usability Scale (SUS) | Immediately after exposure
  Likert scale (5 point) based assessment of software usability. Higher scores on a scale of 1 to 5 represent a better software system usability.
Modified Simulation Effectiveness Tool (SET-M) | Immediately after exposure
  likert scale (3 point) validated assessment of learning satisfaction tool
Time required to complete critical crisis related tasks | 30 days post exposure
  Measured time until critical scenario management events occur
anaphylaxis knowledge test | 30 days post exposure
  validated multiple choice quiz of anaphylaxis knowledge developed by allergists for use with the same curriculum included in our study

CONTACTS AND LOCATIONS:
Overall Officials: Julian Wiegelmann, Dr., Principal Investigator — Sunnybrook Health Science Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
For confidentiality purpose, Participants personal information will not be shared, and any study data that will be sent outside of the research institution will be encrypted by an ID code for each participant.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will become available only after publication in a Peer reviewed medical journal and will follow the paper's policy regarding the specific limit time to remain public.
Access Criteria: After publication

DOCUMENTS (1):
  • Study Protocol (2025-01-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT05729802/Prot_001.pdf